CLINICAL TRIAL: NCT05357430
Title: The Application of Remazolam in Gastroenteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Wang wanxia, Junior Investigator, Yangzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-YKL12-23
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Gastroenterology
Keywords: Remimazolam
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group D1(males) (Experimental): Administration of 0.3μg/kg of remifentanil in advance, then corresponding dose of remimazolam, according to the experimental results of the previous patient.
  Interventions: Drug: Remimazolam
- group D2(females) (Experimental): Administration of 0.3μg/kg of remifentanil in advance, then corresponding dose of remimazolam, according to the experimental results of the previous patient.
  Interventions: Drug: Remimazolam
- group R (Experimental): Administration of 0.3μg/kg of remifentanil in advance, then the calculated dose of remimazolam, according to the experimental results of the previous patient.
  Interventions: Drug: Remimazolam
- group C (Experimental): Administration of 0.3μg/kg of remifentanil in advance, then 1.5-2mg/kg propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — 0.3μg/kg of remifentanil was injected slowly in advance, then different doses of Remimazolam was injected to two groups of D1 and D2, according to up-and-down method.
  Arms: group D1(males); group D2(females)
Drug: Remimazolam — 0.3μg/kg of remifentanil was injected slowly in advance, then the calculated dose from groups of D1 and D2 of remimazolam was injected to group R.
  Arms: group R
Drug: Propofol — 0.3μg/kg of remifentanil was injected slowly in advance, then 1.5-2mg/kg of Propofol was injected to group C
  Arms: group C

SUMMARY:
OBJECTIVE: To study the safety, efficacy and clinical significance of remimazolam in the diagnosis and treatment of patients with daytime gastrointestinal endoscopy, calculate the optimal dose, and conduct relevant verification. Provide a safer and more effective anesthesia solution for the growing special population.

METHODS：Around 160 patients were selected to receive painless gastroenteroscopy.，they were divided into four groups of D1, D2, R and C. Group D1 and D2(including 60 patients) were used to calculate the ED50 and ED95 of the drug. According to up-and-down method, they were slowly injected 0.3μg/kg of remifentanil in advance, then 0.20mg/kg of remimazolam, and gastroscopy was performed after MOAA/S score ≤３. The next patient would be increased 0.05mg/kg of remimazolam if there is a positive standrd, otherwise it would be decreased 0.05mg/kg. And the study was terminated when seven crossing points occurred. One hundred patients were randomly divided into two groups of R and C.Before administration of remimazolam, remifentanil injection 0.3 μg/kg were given intravenously in two groups, respectively (injection rate was 30 s).Then group R was given the calculated dose of remimazolam, and group C was given propofol 1.5-2mg/kg.The success rate of sedation, changes in vital signs, adverse reactions, and postoperative recovery were recorded in the two groups.

DETAILED DESCRIPTION:
The study used up-and-down methods to calculate the ED50 and ED95. According to up-and-down method, group D1 and D2 were slowly injected 0.5μg/kg of remifentanil in advance, then 0.20mg/kg of remimazolam, and gastroscopy was performed after MOAA/S score ≤３. The standard for a positive response in patients undergoing gastroscopy: coughing, swallowing, frowning, and physical movement affecting the operation during the examination. The next patient would be increased 0.05mg/kg of remimazolam if there is a positive standrd, otherwise it would be decreased 0.05mg/kg.And the study was terminated when seven crossing points occurred. Probit regression analysis method was used to calculate the ED50, ED95 and 95%CI of remimazolam combined with remifentanil in painless gastroenteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old; ASA classification I-II grade

Exclusion Criteria:

* Asthma; allergic to the drugs involved and contraindicated; patients with severe respiratory system, cardiovascular system diseases and coagulation insufficiency of liver and kidney function; patients with severe neuropsychiatric system diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Success rate of sedation | 1-3minutes
  After the administration of remimazolam, observe and record the response
Blood pressure value | 1-30minutes
  record the blood pressure before and after administration
Heart rate | 1-30minutes
  record the heart rate before and after administration

SECONDARY OUTCOMES:
Incidence of adverse reactions | 1-30minutes
  Incidence of adverse reactions such as intraoperative movement, choking, respiratory depression, hiccups, nausea and vomiting, dizziness, laryngospasm

CONTACTS AND LOCATIONS:
Overall Officials: Liu M Yu, Director, Principal Investigator — Yangzhou University
Locations (1):
- Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China